CLINICAL TRIAL: NCT01969435
Title: A Phase II Study of Melphalan HCl for Injection (Propylene Glycol-free), Combined With Carmustine, Etoposide, and Cytarabine (BEAM Regimen) for Myeloablative Conditioning in Lymphoma Patients Undergoing Autologous Stem Cell Transplantation
Brief Title: Study of Melphalan HCl for Injection (Propylene Glycol-free), Carmustine, Etoposide, Cytarabine (BEAM Regimen) and Autologous Stem Cell Transplantation for Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201312115
Record Dates: First submitted 2013-10-16; First posted 2013-10-25 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Hodgkin Disease; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Carmustine; etoposide phosphate; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Melphalan, carmustine, etoposide, cytarabine (BEAM) (Experimental): * Day -7, carmustine intravenous (IV) infusion
  * Days -6, -5, -4, and -3, etoposide and cytarabine (IV) infusions twice a day
  * Day -2, melphalan HCl (propylene glycol-free)(IV) infusion
  * Day 0, stem cell transplant.
  Interventions: Drug: Carmustine; Drug: Etoposide phosphate; Drug: Cytarabine; Drug: Melphalan HCl (propylene glycol-free)

INTERVENTIONS:
Drug: Carmustine
  Other Names: BCNU; BiCNU®
Drug: Etoposide phosphate
  Other Names: VP-16; Vepesid
Drug: Cytarabine
  Other Names: Cytosar-U ®; 1-β-Arabinofuranosylcytosine; Arabinosylcytosine; Cytosine arabinoside; Ara-C
Drug: Melphalan HCl (propylene glycol-free)

SUMMARY:
Phase II study is being conducted to confirm the safety and efficacy of high-dose Melphalan HCl for Injection (Propylene Glycol-Free) when included in the BEAM regimen for myeloablative conditioning in lymphoma patients undergoing ASCT

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hodgkin lymphoma or non-Hodgkin lymphoma.
* Eligible for autologous stem cell transplantation.
* 18 to 75 years of age at time of enrollment.
* Adequate autologous graft, defined as an unmanipulated, cryopreserved, peripheral blood stem cell graft containing at least 2 x 10^6 CD34+ cells/kg based on patient body weight
* ECOG performance status ≤ 2
* Normal organ function as defined below:

  * Creatinine clearance > 40 ml/min
  * Total bilirubin ≤2.0 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * LVEF > 40% (by ECHO or MUGA)
  * FEV1 > 50% of predicted and DLCO > or = 50% of predicted
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any other experimental therapy or has received any other experimental therapy within the 4 weeks prior to enrollment.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to melphalan HCl for injection (propylene glycol-free), Captisol, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding women. Women of childbearing potential must have a negative serum pregnancy test within 14 days of study entry.
* Known HIV-positivity. These patients are excluded because of the potential for pharmacokinetic interactions with the study regimen and their antiretroviral therapy and because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 51 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 50
Diagnosis [Number; unit: participants]
  Hodgkin lymphoma | 17
  Diffuse large B-cell lymphoma | 15
  Mantle cell lymphoma | 8
  Other Non-Hodgkin Lymphoma | 10
Remission status prior to autologous stem cell transplant [Number; unit: participants]
  Complete remission | 23
  Partial remission | 25
  Progressive disease | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Toxicity as Measured by Treatment Related Non-hematologic Adverse Events
Description: Adverse events will be assessed using the National Cancer Institute (NCI)-CTCAE version 4.0. Number of events, grade 2 or higher, occurring in 10% or greater of participants. Grade 2 diarrhea and Grade 2 nausea/vomiting were not recorded.
Time Frame: Day -7 through Day 30
Measure: Number; unit: participants
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
participants
  Fever neutropenia | 34
  Fever | 6
  Bacteremia | 7
  Clostridium difficile | 3
  Respiratory infection | 5
  Mucosal infection | 7
  Skin infection | 3
  Genito-urinary tract infection | 3
  Hypotension | 15
  Abdominal pain | 5
  Diarrhea | 8
  Mucositis oral | 27
  Liver enzymes increased | 5
  Bilirubin increased | 5
  Dehydration | 5
  Hyperglycemia | 6
  Hypoalbuminemia | 10
  Hypocalcemia | 12
  Hypokalemia | 14
  Hypophosphatemia | 35
  Pain | 10
  Headache | 7
  Hypoxia | 9
  Rash | 8

2. Primary Outcome: Treatment-related Mortality (TRM)
Description: TRM is defined as death not due to progressive lymphoma prior to Day 100 after transplant
Time Frame: 100 days
Measure: Number; unit: percentage of participants
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
percentage of participants | 0

3. Secondary Outcome: Efficacy as Measured by Response Rates
Description: * The response rates according to each category of response Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD) will be summarized by the proportion of patients meeting each criterion.
  * Evaluated using PET or CT scan and Revised Response Criteria for Malignant Lymphoma
Time Frame: Up to Day 100
Measure: Number; unit: percentage of participants
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
percentage of participants
  Complete response | 84
  Partial response | 4
  Stable disease | 0
  Progressive disease | 12

4. Secondary Outcome: Disease-free Survival
Description: Percentage of patients who survive without any signs or symptoms of cancer at 1 year.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
percentage of participants | 70 [58 to 85]

5. Secondary Outcome: Disease-free Survival
Description: Percentage of patients who survive without any signs or symptoms of cancer at 2 years.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
percentage of participants | 64

6. Secondary Outcome: Time to Engraftment (Neutrophil)
Description: Time from the date of the transplant to the date of neutrophil engraftment.
Time Frame: Assessed up to day 30
Measure: Median (Full Range); unit: days
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
days | 10 [9 to 13]

7. Secondary Outcome: Time to Engraftment (Platelet)
Description: Time from the date of transplant to the date of platelet engraftment.
Time Frame: Assessed up to day 100
Population: One patient did not have platelet engraftment by Day 100
Measure: Median (Full Range); unit: days
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 49
days | 19 [12 to 90]

8. Post Hoc Outcome: Progression-free Survival (PFS) Rate
Description: PFS - Time from start of treatment to the time of progression or death, whichever occurs first.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
percentage of participants | 84 [74 to 95]

9. Post Hoc Outcome: Progression-free Survival Rate (PFS)
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
percentage of participants | 70 [58 to 85]

10. Post Hoc Outcome: Relapse Free Survival
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
percentage of participants | 0

11. Post Hoc Outcome: Overall Survival (OS) Rate
Time Frame: Median follow-up 15.4 months (range 4.7-24.6)
Measure: Number; unit: percentage of participants
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Number analyzed (Participants) | 50
percentage of participants | 10

ADVERSE EVENTS:
Time Frame: Reportable adverse events were collected from the first dose of study treatment (Day -7) through the Day +30 visit.
Description: Reportable adverse events are events grade 2 or higher. Hematologic adverse events are expected and therefore the following adverse events were not collected/reported regardless of grade: anemia, white blood cell decreased, neutrophil count decreased, lymphocyte count decreased, and platelet count decreased. In addition, the following grade 2 non-hematologic adverse events were expected and not collected/reported: nausea, vomiting, diarrhea, anorexia, fatigue, and alopecia.
Arm/Group | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM)
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM) (N=50)
Multi-organ failure due to sepsis (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melphalan, Carmustine, Etoposide, Cytarabine (BEAM) (N=50)
Abdominal pain (Gastrointestinal disorders) | 5
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Allergic reaction (Immune system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Aspartate aminotransferase increased (Investigations) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
BCNU pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blood bilirubin increased (Investigations) | 5
Blood-Coagulase-negative staphylococcus (Infections and infestations) | 3
Blood-Enterobacter clocae/streptococcus mitis (Infections and infestations) | 1
Blood-Klebsiella pneumoniae (Infections and infestations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Catheter related infection (Infections and infestations) | 1
Chills (General disorders) | 2
Clostridium difficile (Infections and infestations) | 3
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Diarrhea (Gastrointestinal disorders) | 8
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 3
Esophageal spasm (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Febrile neutropenia (Infections and infestations) | 34
Fever (General disorders) | 6
Flushing (Vascular disorders) | 2
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
HSV (oral) (Infections and infestations) | 2
Headache (Nervous system disorders) | 7
Heart failure (Cardiac disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 4
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypokalemia (Metabolism and nutrition disorders) | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 35
Hypotension (Vascular disorders) | 15
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9
Ileal obstruction (Gastrointestinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Lethargy (Nervous system disorders) | 1
Localized edema (General disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Mucosal infection (oral candidiasis) (Infections and infestations) | 5
Mucositis oral (Gastrointestinal disorders) | 27
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Non-cardiac chest pain (General disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Parainfluenaza virus type 3 (Infections and infestations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Rectal pain (Gastrointestinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes